CLINICAL TRIAL: NCT00700973
Title: Treating Violence-Prone Substance Use Disorder Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-264
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-02

CONDITIONS: Substance-related Disorders; Violence
Keywords: anger; psychotherapy, brief; diagnosis, dual
MeSH Terms: conditions — Substance-Related Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Substance use disorder usual care
  Interventions: Other: Usual care
- Arm 2 (Experimental): Interpersonal violence prevention intervention
  Interventions: Behavioral: Interpersonal Violence Prevention Intervention

INTERVENTIONS:
Behavioral: Interpersonal Violence Prevention Intervention — This is a cognitive-behavioral approach incorporating cognitive restructuring and behavioral change.
  Arms: Arm 2
Other: Usual care — Substance use disorder usual care
  Arms: Arm 1

SUMMARY:
This project is intended to help substance use disorder patients who perpetrate interpersonal violence against other adults.

DETAILED DESCRIPTION:
Background:

Interpersonal violence (IPV) among substance use disorder (SUD) patients is common, undertreated, and costly. SUD patients have high rates of perpetrating IPV, and IPV is a risk factor for poor response to SUD treatment. Failure to address IPV among SUD patients interferes with treatment effectiveness and contributes to relapse and higher rates of health services use. Nonetheless, SUD treatment programs typically do not include violence prevention interventions and few studies have examined interventions designed to prevent violence perpetration among SUD patients.

Objectives:

This trial evaluated the effectiveness of an IPV-prevention (IPV-P) intervention among patients entering VA SUD treatment who had perpetrated violence in the past year against another adult. Primary objectives were to test the hypotheses that, compared to patients assigned to a control condition (CC), those assigned to IPV-P would (1) improve more on violence and SUD outcomes, and (2) use fewer VA mental health and medical care services, thereby saving costs for VA. Secondary objectives were to test the hypothesis that, compared to patients assigned to CC, those assigned to IPV-P would improve more on legal and alienation problems and social resources.

Methods:

Patients entering VA SUD treatment who met eligibility criteria (past-year violence; cognitively intact) and provided informed consent were assigned to SUD usual care plus either a CC (N=60) or IPV-P (N=59) intervention using a recurrent institutional design. That is, the IPV-P and CC conditions were run in alternate 3-month periods. The manualized IPV-P group intervention, based on a Cognitive-Behavioral approach, consisted of 8 in-person group sessions over 1 month, followed by telephone calls once a month for 3 months. The manualized CC was designed to control for non-specific treatment effects associated with the IPV-P condition, i.e., counselor time and attention, peer support, patients' expectations that additional sessions provide benefit. It consisted of 8 in-person group sessions over 1 month that reviewed material covered in usual SUD treatment, but with novel methods used to deliver the IPV-P intervention (role-play, homework, group activities). CC included the booster telephone sessions (once per month for 3 months). Participants were assessed at baseline and end-of-intervention (4 months post-baseline) and 6 and 12 months post-intervention (i.e., 10 and 16 months post-baseline) for primary and secondary outcomes and non-VA healthcare. Assessments consisted of the Addiction Severity Index (ASI, to assess Alcohol, Drugs, Psychiatric, and Legal functioning), the Conflicts Tactics Scale (CTS, to assess Psychological Aggression and Physical Assault against another adult), the Multidimensional Personality Questionnaire (MDQ, to assess Alienation, Stress Reaction, and Aggression), and the Life Stressors and Social Resources Inventory (LISRES, to assess family and friends resources). VA health care is being assessed with VA databases. Response rates at 4, 10, and 16 months were 90%, 79%, and 73%, respectively, and did not differ between the IPV-P and CC groups. Follow-up analyses compared the IPV-P to the CC group on outcomes using analyses of covariance that controlled for the baseline value of the outcome.

Status:

We are still completing portions of this project: (1) conducting mixed effects regression analyses to compare the CC and IPV-P groups on primary and secondary outcomes (these analyses are partially completed), and (2) using data on VA health care utilization to compare the two groups on VA health care costs (permission to download these data has been obtained, and we are working with HERC investigators to download and analyze the data).

ELIGIBILITY:
Inclusion Criteria:

* Entering VA substance use disorder treatment
* past-year violence
* cognitively intact

Exclusion Criteria:

* Not entering VA substance use disorder treatment
* no past-year violence
* cognitively not intact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Timko, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

REFERENCES:
- [Result] Timko C, Desai A, Blonigen DM, Moos BS, Moos RH. Driving while intoxicated among individuals initially untreated for alcohol use disorders: one- and sixteen-year follow-ups. J Stud Alcohol Drugs. 2011 Mar;72(2):173-84. doi: 10.15288/jsad.2011.72.173. PMID 21388590
- [Result] Blonigen DM, Timko C, Moos BS, Moos RH. Impulsivity is an independent predictor of 15-year mortality risk among individuals seeking help for alcohol-related problems. Alcohol Clin Exp Res. 2011 Nov;35(11):2082-92. doi: 10.1111/j.1530-0277.2011.01560.x. Epub 2011 Jun 1. PMID 21631544
- [Result] Makin-Byrd K, Cronkite RC, Timko C. The influence of abuse victimization on attendance and involvement in mutual-help groups among dually diagnosed male veterans. J Subst Abuse Treat. 2011 Jul;41(1):78-87. doi: 10.1016/j.jsat.2011.02.001. Epub 2011 Mar 10. PMID 21396794
- [Result] Timko C, Sutkowi A, Cronkite RC, Makin-Byrd K, Moos RH. Intensive referral to 12-step dual-focused mutual-help groups. Drug Alcohol Depend. 2011 Nov 1;118(2-3):194-201. doi: 10.1016/j.drugalcdep.2011.03.019. Epub 2011 Apr 22. PMID 21515004

RESULTS

PARTICIPANT FLOW:
Groups:
- IPV-P: Interpersonal violence prevention intervention
  Interpersonal Violence Prevention Intervention: This is a cognitive-behavioral approach incorporating cognitive restructuring and behavioral change.
Period: Overall Study
Arm/Group | Usual Care | IPV-P
Started | 71 | 70
Completed | 63 | 63
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 71 | 70 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8) | 51 (8) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 71 | 70 | 141
Race/Ethnicity, Customized [Number; unit: participants]
  White | 34 | 34 | 68
  Non-White | 37 | 36 | 73
Region of Enrollment [Number; unit: participants]
  United States | 71 | 70 | 141

OUTCOME MEASURES:

1. Primary Outcome: Addiction Severity Index Legal Composite
Description: Scores range from 0 to 1, with higher scores indicating more severe legal problems.
Time Frame: One year post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 68 | 68
units on a scale | .038 (.049) | .012 (.049)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/70
Other Adverse Events (participants affected / at risk) | 0/71 | 0/70

LIMITATIONS AND CAVEATS:
A limitation of the trial (not a result or conclusion) is that high proportions of patients reported abstinence at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes